CLINICAL TRIAL: NCT02409537
Title: Cardiovascular Risk and Benefits From Antioxidant Dietary Intervention With Red Wine in Asymptomatic Hypercholesterolemics
Brief Title: Effects of Dietary Antioxidants to Prevent Cardiovascular Disease
Acronym: RWTAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeromedical Center, Thessaloniki (Other)
Responsible Party: Principal Investigator, Christina Apostolidou, Aristotle University of Thessaloniki, School of engineering, Faculty of Chemical Engineering, Division of technology laboratory of food and process engineering, Aeromedical Center, Thessaloniki
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0011
Record Dates: First submitted 2015-03-29; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia; Healthy
Keywords: Asymptomatic hypercholesterolemia,; cardiovascular risk,; total antioxidant capacity; red wine polyphenol content; vitamin E.; resveratrol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non cholesterolemic individuals (Active Comparator): Individuals with normal cholesterol levels will consume red wine for 1 month. There will be 1 month of wash out period. After 1 month of wash out period resveratrol will be consumed for 1 month and finally after 1 month wash out period placebo will be administered for 1 month.
  Interventions: Dietary Supplement: red wine; Dietary Supplement: resveratrol; Other: placebo
- Asymptomatic Hypercholesterolemics (Active Comparator): individuals with high levels of cholesterol with no cardiovascular disease Those individuals will consume red wine for 1 month. There will be 1 month of wash out period. After 1 month of wash out period resveratrol will be consumed for 1 month and finally after 1 month wash out period placebo will be administered for 1 month.
  Interventions: Dietary Supplement: red wine; Dietary Supplement: resveratrol; Other: placebo

INTERVENTIONS:
Dietary Supplement: red wine — the individuals were given red wine to consume for 1 month then a wash out period of 1 month
Dietary Supplement: resveratrol — the individuals were given resveratrol for 1 month and then 1 month wash out period
Other: placebo — the individuals were given placebo for 1 month

SUMMARY:
Background & Aims: The role of red wine in cardiovascular risk prevention has been documented by several epidemiological studies in patients and normocholesterolemic healthy individuals. However, it is unclear whether hypercholesterolemic individuals free of cardiovascular disease would equally benefit from moderate red wine consumption to prevent atherosclerosis and the development of cardiovascular disease.

Methods: Forty (40) healthy volunteers males and females were recruited, divided into 2 age-adjusted groups according to their total cholesterol levels; in asymptomatic hypercholesterolemics (AHC ), and normocholesterolemics (NC ). Total Antioxidant Capacity (TAC ), Lipid profile, Vitamin E, and cardiovascular risk indexes ( LDL /HDL and Vitamin E/TC ) were evaluated in the blood serum of all subjects prior to and 1 month after once daily red wine consumption as well as prior to and after being given a placebo drink following a 1 month wash out period and resveratrol for 1 month after wash out period..

DETAILED DESCRIPTION:
Study design and measurements This study is a cross-over field trial. Participants were asked to consume a specific variety of red wine "tannat" daily in their diet for one month. After a wash-out period of one month, the same participants were asked to consume a placebo drink daily for another month. Quantitative measurements of blood lipids, vitamin E, and Total Antioxidant Capacity before and after consumption of wine and placebo were measured. The study aimed to investigate whether consumption of red wine is associated with any changes in the levels of blood lipids, vitamin E, and Total Antioxidant Capacity and whether such changes - if any -equally occur in hypercholesterolemic individuals.

Participants were advised to abstain from consuming antioxidant supplements, antioxidant-rich foods (including deep-colored fruits and vegetables such as berries, tomatoes, carrots, broccoli, apples and plums, green tea, caffeine and chocolate), caffeine and alcohol 2 weeks prior to the beginning of initial measurements and during the 3-month experimental period. Participants (occasional alcohol drinkers) included in the study received no monetary compensation. According to the U.S. Department of Agriculture 2010 Dietary Guidelines, moderate drinking corresponds to one drink per day for women and two for men14. Consequently, female subjects were given 5 bottles of red wine for 1 month (1 glass per day), and male subjects were given 10 bottles (2 glasses/per day) and instructed to report any side effects or failure to participate. The single grape variety of Tannat, from a location in Northern Greece, was selected among several varieties of red wine for its content in phenolic compounds and high antioxidant gradient when tested in vitro. Participants were encouraged to not alter their dietary habits or physical activity level during the study. To verify their compliance with the instructions provided, we interviewed them before and after the experiment, and we also measured the quantity of wine used. One day prior to the beginning of the intervention, participants underwent physical and routine biochemical examinations and completed two questionnaires, one related to their health status and the other to their characteristics. To confirm protocol adherence, a team of colleagues contacted the participants by telephone every 2nd day and they visited the clinic to obtain 1 bottle of wine and answered a questionnaire regarding their adherence with the protocol requirements.

For each subject, measurements of serum TAC and vitamin E were performed pre and post 1 month of red wine ingestion and pre and post placebo drink ingestion after a 1 month wash out period. For vitamin E measurements, fasting subjects were requested to abstain from alcohol for 24 hours prior to the blood draw. Serum levels of Total Cholesterol (TC), triglycerides (TG), HDL-cholesterol, and LDL-cholesterol were also measured by enzymatic methods. For serum HDL-cholesterol levels, fasting blood was collected in tubes with a clot activator and was determined enzymatically.

For the assessment of cardiovascular risk, pre and post red wine consumption ratios (LDL/HDL-cholesterol and vitamin E/TC) were calculated. TG/HDL-cholesterol, a marker for insulin resistance, was also proposed as a surrogate marker of cardiovascular risk assessment. TC/HDL and LDL/HDL are also considered to be strong predictors of the degree of clinical benefit from lipid-lowering interventions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with normal or high cholesterol level with no cardiovascular disease

Exclusion Criteria:

* documented dyslipidemia (abnormal level of fat or cholesterol (very high or very low),
* chronic liver disease, malnutrition, neoplastic or acute infectious diseases,
* habitual use of vitamin supplements.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Total antioxidant activity (TAC) | 6 months
  TAC was measured after 1 month of red wine consumption, resveratrol and placebo and wash out periods in between
Vitamin E | 6 months
  Vitamin E was measured after 1 month of red wine consumption, resveratrol and placebo and wash out periods in between
Total Cholesterol | 6 months
  Total cholesterol was measured after 1 month of red wine consumption, resveratrol and placebo and wash out periods in between
LDL/HDL | 6 months
  The ratio LDL/HDL was measured after 1 month of red wine consumption, resveratrol and placebo and wash out periods in between

SECONDARY OUTCOMES:
Vitamin E/ Total Cholesterol | 6 months
  The ratio Vitamin E/ Total Cholesterol was measured after 1 month of red wine consumption, resveratrol and placebo and wash out periods in between

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Adamopoulos, PhD, Study Director — Aristotle University of Thessaloniki, School of engineering, Faculty of Chemical Engineering, Division of technology laboratory of food and process engineering,; Christina Apostolidou, MS, Principal Investigator — Aristotle University of Thessaloniki, School of engineering, Faculty of Chemical Engineering, Division of technology laboratory of food and process engineering,

REFERENCES:
- [Result] Quinones M, Miguel M, Aleixandre A. Beneficial effects of polyphenols on cardiovascular disease. Pharmacol Res. 2013 Feb;68(1):125-31. doi: 10.1016/j.phrs.2012.10.018. Epub 2012 Nov 19. PMID 23174266
- [Result] Zenebe W, Pechanova O, Bernatova I. Protective effects of red wine polyphenolic compounds on the cardiovascular system. Exp Clin Cardiol. 2001 Fall;6(3):153-8. PMID 20428452
- [Result] Roerecke M, Rehm J. Chronic heavy drinking and ischaemic heart disease: a systematic review and meta-analysis. Open Heart. 2014 Aug 6;1(1):e000135. doi: 10.1136/openhrt-2014-000135. eCollection 2014. PMID 25332827